CLINICAL TRIAL: NCT07286110
Title: Effect of Chinese Herbal Intervention (Qiqi Shengmai Formula) for Moyamoya Vasculopathy in Cerebral Hemodynamics (CHIMES ): a Single-center, Prospective, Randomized Controlled Study
Brief Title: Chinese Herbal Therapy (Qiqi Shengmai Formula) for Moyamoya Vasculopathy: The CHIMES Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ziyang He, Sub-Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShanghaiZhongshan
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Moyamoya Disease; Moyamoya Syndrome
MeSH Terms: conditions — Moyamoya Disease | interventions — Medicine, Chinese Traditional; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Traditional Chinese and Conventional Medical Treatment Group (Experimental): Conventional Medical Treatment:
  For ischemic-type moyamoya disease, antiplatelet monotherapy with cilostazol is administered, while antiplatelet therapy is not recommended for asymptomatic patients or those with hemorrhagic-type moyamoya disease. For patients with concomitant dyslipidemia, statins and evolocumab may be added, with low-density lipoprotein cholesterol controlled to 70 mg/dL (1.8 mmol/L). Blood pressure is maintained at 140/90 mmHg, and glycemic management targets a hemoglobin A1c level of <7.0%.
  Traditional Chinese Medicine (TCM) Treatment:
  Patients receive the standardized TCM formula Qiqi Shengmai Decoction (composed of Astragali Radix, Rehmanniae Radix Praeparata, Schisandrae Fructus, Bupleuri Radix, Paeoniae Radix Alba, and Notoginseng Radix). The prescription is taken twice daily, one dose per administration, for six consecutive weeks, with each dose consumed 30 minutes after breakfast and dinner
  Interventions: Drug: Traditional Chinese Medicine (TCM) Treatment; Drug: Conventional medical treatment
- Conventional Medical -Only Treatment Group (Placebo Comparator): Conventional Medical Treatment： For ischemic-type moyamoya disease, antiplatelet monotherapy with cilostazol is administered, whereas antiplatelet therapy is not recommended for asymptomatic patients or those with hemorrhagic-type moyamoya disease. For patients with concomitant dyslipidemia, statins and evolocumab may be added, with low-density lipoprotein cholesterol controlled to 70 mg/dL (1.8 mmol/L). Blood pressure is maintained at 140/90 mmHg, and glycemic management targets a hemoglobin A1c level of <7.0%.
  TCM Placebo:
  The placebo consists primarily of medicinal starch, food-grade caramel coloring (for color correction), and a bittering agent (for flavor adjustment). Its appearance-including shape, size, color, and taste-is identical to that of the herbal preparation. It is administered twice daily, one dose at each administration, for six consecutive weeks, taken 30 minutes after breakfast and dinner.
  Interventions: Drug: Conventional medical treatment; Drug: TCM Placebo

INTERVENTIONS:
Drug: Traditional Chinese Medicine (TCM) Treatment — Patients receive the standardized TCM formula Qiqi Shengmai Decoction (composed of Astragali Radix, Rehmanniae Radix Praeparata, Schisandrae Fructus, Bupleuri Radix, Paeoniae Radix Alba, and Notoginseng Radix). The prescription is taken twice daily, one dose per administration, for six consecutive weeks, with each dose consumed 30 minutes after breakfast and dinner
  Arms: Integrated Traditional Chinese and Conventional Medical Treatment Group
Drug: Conventional medical treatment — For ischemic-type moyamoya disease, antiplatelet monotherapy with cilostazol is administered, while antiplatelet therapy is not recommended for asymptomatic patients or those with hemorrhagic-type moyamoya disease. For patients with concomitant dyslipidemia, statins and evolocumab may be added, with low-density lipoprotein cholesterol controlled to 70 mg/dL (1.8 mmol/L). Blood pressure is maintained at 140/90 mmHg, and glycemic management targets a hemoglobin A1c level of <7.0%.
Drug: TCM Placebo — The placebo consists primarily of medicinal starch, food-grade caramel coloring (for color correction), and a bittering agent (for flavor adjustment). Its appearance-including shape, size, color, and taste-is identical to that of the herbal preparation. It is administered twice daily, one dose at each administration, for six consecutive weeks, taken 30 minutes after breakfast and dinner.
  Arms: Conventional Medical -Only Treatment Group

SUMMARY:
Patients diagnosed with moyamoya vasculopathy by imaging and classified as having the Traditional Chinese Medicine (TCM) syndrome of liver-yang hyperactivity will be enrolled. On the basis of standardized Western medical management, participants will receive the standardized TCM herbal formula "Qiqi Shengmai Formula" (comprising Astragali Radix, Rehmanniae Radix Praeparata, Schisandrae Fructus, Bupleuri Radix, Paeoniae Radix Alba, and Notoginseng Radix). Structured follow-up will be conducted. By comparing endpoint indicators across different treatment regimens, the study aims to evaluate the efficacy of integrated TCM-Western medicine therapy for moyamoya vasculopathy and to generate evidence-based support for an integrated diagnostic and therapeutic model.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging findings meeting the Western medical diagnostic criteria for moyamoya vasculopathy
2. Age between 18 and 80 years
3. The patient and family members are fully informed and voluntarily consent to participation, with the informed consent process conducted in accordance with GCP requirements
4. Willingness to receive Traditional Chinese Medicine treatment
5. Traditional Chinese Medicine syndrome differentiation consistent with liver-yang hyperactivity

Exclusion Criteria:

1. Acute cerebrovascular events within the preceding 6 weeks
2. Known allergy to contrast agents or to the investigational medication
3. Presence of severe primary diseases involving the cardiac, pulmonary, hepatic, renal, endocrine, or hematopoietic systems
4. Pregnant or breastfeeding women
5. Patients scheduled to undergo cerebral revascularization surgery
6. Participation in other ongoing clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
CT Perfusion | Baseline, at 3 months, 6 months, and 12 months after enrollment
  Cerebral perfusion parameters measured by CT perfusion imaging, including cerebral blood flow (CBF), cerebral blood volume (CBV), mean transit time (MTT), and time to peak (TTP), to evaluate cerebral hemodynamics.

SECONDARY OUTCOMES:
Digital Subtraction Angiography | Baseline, 12 months after enrollment
  Cerebral angiographic characteristics assessed by digital subtraction angiography, including degree of arterial stenosis/occlusion, collateral vessel formation, and Suzuki stage.
Integrated Head-Neck High-Resolution Vessel Wall MRI | Baseline, 6 months, and 12 months after enrollment
  Intracranial arterial wall characteristics assessed by high-resolution vessel wall MRI, including vessel wall thickening, enhancement pattern, and lumen diameter.
TCM Symptom Scale | Baseline, at 3 months, 6 months, and 12 months after enrollment
  Traditional Chinese Medicine symptom severity assessed using a standardized TCM Symptom Scale.
  Total score ranges from 0 to 45, with higher scores indicating more severe symptoms.
Modified Rankin Scale (mRS) | Baseline, at 3 month, 6 months, and 12 months after enrollment
  Functional outcome assessed by the Modified Rankin Scale, ranging from 0 to 6, where higher scores indicate worse functional outcome.
TCM Constitution Classification | Baseline, at 3 month, 6 month, and 12 months after enrollment
  Traditional Chinese Medicine constitution type assessed using a standardized TCM Constitution Classification questionnaire, categorizing participants into predefined constitution types.
Montreal Cognitive Assessment (MoCA) | Baseline, and at 3, 6, and 12 months after enrollment
  Cognitive function assessed by the Montreal Cognitive Assessment, with total scores ranging from 0 to 30, where higher scores indicate better cognitive function.
National Institutes of Health Stroke Scale (NIHSS) | Baseline and at 3, 6, and 12 months after enrollment
  Neurological deficit severity assessed by the National Institutes of Health Stroke Scale, with scores ranging from 0 to 42, where higher scores indicate more severe neurological deficits.

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Xuhui District, Shanghai 200032,China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No